CLINICAL TRIAL: NCT07314008
Title: Comparison of Left Bundle Branch Area Pacing and Minimized Ventricular Pacing in Patients With Sinus Node Dysfunction and Atrioventricular Conduction Delay: A Multicenter, Randomized Controlled Clinical Trial
Brief Title: Left Bundle Branch Versus Minimized Ventricular Pacing in Patients With Sick Sinus Syndrome and Prolonged AV Interval
Acronym: CLOSE-AV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Severance Hospital (Other); Samsung Medical Center (Other); Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Gi-Byoung Nam, professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC2024-0579
Record Dates: First submitted 2025-11-24; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-05

CONDITIONS: Sick Sinus Syndrome; Atrioventricular Nodal Dysfunction
MeSH Terms: conditions — Sick Sinus Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LBBAP (Experimental)
  Interventions: Device: LBBAP
- MVP (Active Comparator)
  Interventions: Device: MVP

INTERVENTIONS:
Device: LBBAP — * All pacemaker implantation should be performed in standard manner.
  * A lead should be placed in the right atrial appendage or septum where acceptable sensing (P wave >1mV) and pacing threshold (<1V at 0.4ms width).
  * V lead should be placed in the right ventricular septum where conduction system pacing can be achieved with acceptable sensing and pacing threshold. The pacing morphology should be compatible with His bundle pacing, right ventricular pacing, selective and non-selective left bundle branch pacing, or left fascicular pacing.
  * The primary objective for the LBBAP group is the achievement of conduction system capture with LBBAP. However, based on the physician's discretion or the situations in the operating room, His bundle pacing can be accepted as alternatives to LBBAP.
  Arms: LBBAP
Device: MVP — * All pacemaker implantation should be performed in standard manner.
  * A lead should be placed in the right atrial appendage or septum where acceptable sensing (P wave >1mV) and pacing threshold (<1V at 0.4ms width).
  * V lead should be placed in the right ventricular apex or septum where acceptable sensing (R wave >5mV) and pacing threshold (<1V at 0.4ms width)
  * The rhythmiQTM mode should be turned on
  * Sensing and pacing AV intervals recommended to be >300ms (default value or more), and should not be <200ms to minimize the ventricular pacing.
  Arms: MVP

SUMMARY:
The goal of this clinical trial is to compare two pacemaker strategies: Left Bundle Branch Area Pacing (LBBAP) and Minimized Ventricular Pacing (MVP) in patients requiring a permanent pacemaker for sick sinus syndrome and prolonged AV interval. It will also evaluate the safety and feasibility of the LBBAP method in these patients.

The main questions it aims to answer is:

*Is LBBAP with physiological AV interval better than Minimized Ventricular Pacing?

Researchers will compare the LBBAP group (aiming for conduction system capture with physiological AV intervals) to the MVP group (aiming to minimize ventricular pacing with prolonged AV intervals) to evaluate the optimal pacing strategy.

Participants will:

* Be randomly assigned to either the LBBAP group or the MVP group.
* Undergo a pacemaker implantation procedure according to the specific criteria for their assigned group.
* Visit the clinic for regular checkups to measure pacing function and ensure the device settings remain compliant with the study protocol.

DETAILED DESCRIPTION:
Eligible subjects who provide written informed consent will be randomly assigned in a 1:1 ratio to either the LBBAP group or the MVP group. Randomization will be available 24 hours a day using an Interactive Web Response System (IWRS). Randomization will be stratified by the presence of a history of AF. For patients who meet the inclusion and exclusion criteria before the procedure, randomization will be performed beforehand. For patients with SSS requiring PPM implantation, whose AV conduction status cannot be evaluated before the procedure due to conditions such as junctional rhythm, marked bradycardia (<50 bpm), or isorhythmic dissociation, randomization can be performed after the demonstration of PR with atrial pacing at a targeted atrial rate of 60 bpm during the procedure.

LBBAP group

* All pacemaker implantation should be performed in a standard manner.
* A lead should be placed in the right atrial appendage or septum where acceptable sensing (P wave >1mV) and pacing threshold (<1V at 0.4ms width) are achieved.
* V lead should be placed in the right ventricular septum where conduction system pacing can be achieved with acceptable sensing and pacing threshold. The pacing morphology should be compatible with His bundle pacing, right ventricular pacing, selective and non-selective left bundle branch pacing, or left fascicular pacing.

LBB pacing -Lead position deep in the interventricular septum, ~1-2cm from the distal His bundle potential, LBB potential to QRS interval in the range of 15-34 ms, normal QRS axis, fulfilled criteria for conduction system capture.

Left fascicular pacing

-Capture of the LBB fascicles or its distal arborization, short potential to QRS interval (<25ms), abnormal paced QRS axis with presence of criteria for conduction system capture. Pacing is more distant from the His bundle (2-4cm), defined as left anterior, mid-septal, and posterior fascicle.

Left ventricular septal pacing)

* Capture of the left side of the interventricular septum without direct activation of the left conduction system.
* Terminal R-wave in V1, deep septal position of the pacing lead in the basal to mid-septal area, absence of criteria for conduction system capture.

The primary objective for the LBBAP group is the achievement of conduction system capture with LBBAP. However, based on the physician's discretion or the situations in the operating room, His bundle pacing can be accepted as alternatives to LBBAP.

MVP group

* All pacemaker implantation should be performed in a standard manner.
* A lead should be placed in the right atrial appendage or septum where acceptable sensing (P wave >1mV) and pacing threshold (<1V at 0.4ms width).
* V lead should be placed in the right ventricular apex or septum where acceptable sensing (R wave >5mV) and pacing threshold (<1V at 0.4ms width).
* The RythmiQ™ mode should be turned on.
* Sensing and pacing AV intervals recommended to be >300ms (default value or more), and should not be <200ms to minimize the ventricular pacing.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Sinus node dysfunction with symptoms
* Atrioventricular conduction delay (PR interval > 200ms)

Exclusion Criteria:

* Subject was unable to provide written informed consent or participate in long-term follow-up.
* Permanent atrial fibrillation
* Pre-existing cardiac implantable electronic device
* Persistent advanced atrioventricular conduction disturbance (2:1 block, Mobitz type II, or 3rd degree)
* Mechanical tricuspid valve
* Ventricular septal defect or scar
* Left ventricular ejection fraction < 35% who indicated cardiac resynchronization therapy
* Previous heart transplantation
* Pregnant and/or lactating women
* Life expectancy <2 year
* Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Rate of composite of all-cause mortality, heart failure hospitalization and persistent atrial fibrillation | 2 years
  * All cases of mortality after randomization will be counted.
  * Worsening heart failure includes heart failure hospitalization or urgent heart failure visit (outpatient or emergency department)
  * Persistent atrial fibrillation is defined when there are at least seven consecutive days with 22 hours of device-recorded AF per day or at least one day with an episode of AF lasting at least 22 hours, which is interrupted by electrical or chemical cardioversion.

SECONDARY OUTCOMES:
- All cause mortality | 2 years
  All cases of mortality after randomization will be counted.
- Ischemic stroke or systemic embolism | 2 years
  Composite of ischemic stroke or systemic embolism during follow-up
Heart failure rehospitalization | 2 years
  * The patient is admitted to the hospital with a primary diagnosis of HF
  * The patient's length-of-stay in hospital extends for at least 24 hours
  * The patient exhibits documented at least one new or worsening symptoms due to HF on presentation
  * The patient has objective evidence of new or worsening HF, consisting of at least two physical examination findings or one physical examination and one laboratory criterion.
  * The patient receives at least one of the following treatments specifically for HF
Any rehospitalization | 2 years
  Any rehospitalization after randomization
Rehospitalization from cardiac cause | 2 years
  Rehospitalization for the deterioration of cardiovascular conditions
Quality of life measurement | 2 years
  Quality of life questionnaire and baseline and 24 months. Quality of life is assessed using: 1) 36-Item Short Form Health Survey (SF-36), and 2) Kansas City Cardiomyopathy Questionnaire-12 (KCCQ-12). Both scales range from 0 to 100, with higher scores indicating better health status.
Incidence of Clinical AF | 2 years
  AF detected on 12-lead or other forms of ECG
Quality of life measurement | 2 years
  Quality of life questionnaire and baseline and 24 months. Quality of life will be assessed using the 36-Item Short Form Health Survey (SF-36). This instrument comprises 36 questions covering 8 health domains. Each domain is scored on a scale from 0 to 100, with higher scores indicating a better quality of life/health status

OTHER OUTCOMES:
Periprocedural complications | Periprocedural
  Complications related to the procedure
Incidence of subclinical AF with pre-specified durations | 2 years
  AF lasting >5min, >1 hour, >6 hours, >1 day, and >7 days
Procedural success | Periprocedural
  Achievement of LBB area pacing (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea